CLINICAL TRIAL: NCT06220461
Title: Folic Acid Supplementation to Reduce the Severity of Anemia and Blood Transfusions in Extremely Preterm Infants
Brief Title: Folic Acid Supplementation to Reduce Anemia in Extremely Preterm Infants
Acronym: FASCINATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB23-1665
Record Dates: First submitted 2024-01-10; First posted 2024-01-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-11

CONDITIONS: Extreme Prematurity; Anemia of Prematurity
Keywords: extreme preterm; folic acid deficiency; anemia of prematurity; neonatal blood transfusion
MeSH Terms: conditions — Anemia; Folic Acid Deficiency | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Oral folic acid 50 mcg daily starts at 14 days of age
  Interventions: Dietary Supplement: Folic acid
- Control (No Intervention): No additional folic acid supplementation

INTERVENTIONS:
Dietary Supplement: Folic acid — Infants allocated to the intervention group will receive folic acid (50 mcg flat dose/day) starting at 14 days of age.
  Arms: Experimental group

SUMMARY:
Anemia of Prematurity (AOP) is very common in extremely preterm infants and often leads to blood transfusions. Folic acid, essential for growth and DNA synthesis, is deficient in premature infants. Despite the adoption of folic acid supplementation, evidence supporting its effectiveness in preventing AOP remains scarce. Recommendations for folic acid intake exceed what's naturally found in breast milk, particularly for extremely low birthweight infants. Practices regarding folic acid supplementation vary widely, prompting the need for research. The FACINATE trial aims to determine if additional folic acid supplementation improves hemoglobin levels and reduces late blood transfusions in extremely preterm infants, a question not addressed in current literature.

DETAILED DESCRIPTION:
Anemia of prematurity (AOP) affects nearly all extremely preterm or extremely low birthweight (ELBW; birthweight <1000 g) infants. AOP's development involves various factors such as exacerbation of newborn physiological anemia, reduced response to erythropoietin after birth, frequent blood sampling, short lifespan of red blood cells, and rapid blood volume increase during growth.

To manage this anemia, most infants receive packed red blood cell transfusions, often based on specific hemoglobin thresholds. Despite efforts to minimize transfusion needs in ELBW infants, over 80% still require transfusions during their initial hospital stay. However, these transfusions come with potential adverse effects like infections, immune imbalances, lung and gut injuries, bronchopulmonary dysplasia, and retinopathy of prematurity.

Folic acid is crucial for fetal and postnatal development, playing a central role in DNA synthesis and supporting cell division. Its deficiency can hinder DNA synthesis, cause erythroblast apoptosis, and lead to anemia due to ineffective erythropoiesis. Preterm infants often lack sufficient folic acid, even more so in unfortified breast milk, which contains lower levels than recommended for adequate intake.

Supplementing folic acid for preterm infants began in the early 1990s based on limited studies on low-birth-weight (LBW) infants, primarily formula-fed and weighing >1000 grams. Despite its widespread use, there's insufficient robust evidence specifying the ideal dosage or confirming its effectiveness in preventing AOP or improving hemoglobin levels.

Unfortified breast milk's folic acid content falls short of recommended levels, especially for ELBW infants due to limited hepatic stores and rapid growth. Fortified breast milk or preterm formulas provide varying amounts of folic acid but might still be insufficient, especially for infants on restricted fluid intake due to lung injury.

The FACINATE trial aims to investigate whether additional supplementation of 50 mcg/day of folic acid improves hemoglobin levels and reduces late (>14 days of age) blood transfusions in extremely preterm infants, a specific question not yet explored in existing literature.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at <29 weeks of gestational age admitted to Foothill Medical Centre.
* Postnatal age 14 days.
* On minimum enteral feeding of 100 mL/kg/day

Exclusion Criteria:

* Infants with major congenital or chromosomal anomalies
* Infants with ongoing pulmonary or gastroenterology hemorrhage by 14 days of life.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | At 34-36 weeks corrected gestational age
  The difference in hemoglobin levels between the two groups

SECONDARY OUTCOMES:
Red blood cell transfusion | After 14 days of age and until 36 weeks corrected gestational age
  Number of required red blood cell transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Belal Alshaikh, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No